CLINICAL TRIAL: NCT06229626
Title: Evaluation of an Intensive Training Program for Patients with Hereditary Spastic Paraparesis SPG4/Spast
Acronym: WALK-up
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP230987
Record Dates: First submitted 2023-12-13; First posted 2024-01-29 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Hereditary Spastic Paraparesis
Keywords: physical rehabilitation program; hereditary spastic paraparesis
MeSH Terms: conditions — Spastic Paraplegia, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the reeducation group (Experimental): The population included in the reeducation group will benefit, in addition to their usual physiotherapy care (at least 1 session per week), from :
  * 1 group physiotherapy session per week at the ICM or by videoconference from home for 6 weeks
  * 2 sessions per week at home with video support sent by e-mail for 6 weeks
  These 3 additional video or group sessions will last 30 min. These sessions will be created and adjusted by a physiotherapist and a Physical and Rehabilitation Medicine doctor. They will include exercises such as :
  * Stretching
  * posture
  * Muscle strengthening
  * Proprioception
  And will be performed in standing, sitting and lying positions.
  Interventions: Other: intensive reeducation
- The control group (No Intervention): usual physiotherapy care (at least 1 session per week)

INTERVENTIONS:
Other: intensive reeducation — * 1 group physiotherapy session per week at the ICM or by videoconference from home for 6 weeks
  * 2 sessions per week at home with video support sent by e-mail for 6 weeks
  Arms: the reeducation group

SUMMARY:
Hereditary spastic paraparesis is a group of inherited neurological diseases. Only symptomatic treatments exist for the moment. The Modifspa study (cf citation) carried out by the team showed that patients perceived a feeling of effectiveness of physiotherapy on lower limb spasticity. The aim of the Walk-up study is to objectivize this feeling of efficacy on gait disorders in these patients.

This is an interventional study using physical training. The study is prospective, open, randomized in 2 parallel groups, one of which is a control group. Analyses will be comparative between the 2 groups during the course of the study.

DETAILED DESCRIPTION:
Following an initial study carried out by the team (cf citation), physiotherapy appeared to be the most useful therapy for coping with spasticity, particularly when practised at least 3 times a week. The hypothesis is that this feeling experienced by patients is accurate, and that more frequent physiotherapy (3 additional sessions/week) significantly improves patients' walking speed, with a functional objective.

The main aim of the WALK-UP study is to evaluate the efficacy of a 6-week intensive physical rehabilitation program on walking speed in patients with SPG4 / SPAST-HSP. This is the most frequent genotype in Hereditary Spastic Paraparesis. All patients included in the study will receive at least one physiotherapy session per week in a liberal practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient with molecular diagnosis of hereditary spastic paraparesis based on pathogenic variant of SPAST gene,
* Walking possible for 6 minutes without human assistance (one or more technical aids are authorized: e.g. cane, walker, orthoses),
* At least 1 physiotherapy session per week already in place.
* Understanding of the protocol
* Possibility of connecting to the Internet from home to access video material provided as part of the protocol.

Exclusion Criteria:

* Botulinum toxin injection within 2 months of protocol inclusion
* Discontinuation of private physiotherapy,
* Refusal to participate in the protocol,
* Participation in another interventional clinical trial evaluating a health product or in a randomized clinical trial
* Pregnant women
* Not affiliated to a social security scheme or beneficiary of such a scheme
* Patient under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
to compare the before-and-after variation in distance covered in 6 minutes between the intensive physical rehabilitation group and the control group. | 6 weeks
  6-minute walk test carried out in the presence of a clinician trained in this test. The patient walks for 6 minutes on a circuit of known distance, identical for each patient. The clinician times the walking time and measures the distance covered during 6 minutes. This test is performed at inclusion and again at 6 weeks

SECONDARY OUTCOMES:
compare the before-after variation in distance covered in 6 minutes | 18 weeks
  6-minute walk test carried out in the presence of a clinician trained in this test. This test is performed at inclusion and again at 18 weeks
compare the before-after variation in walking speed over a 10-meters test | 18 weeks
  10-meters test carried out in the presence of a clinician trained in this test. This test is performed at inclusion and again at 18 weeks
compare the clinical evolution of spasticity | 18 weeks
  clinical evolution of spasticity using Spastic Paraplegia Rating Scale (SPRS)
compare the lower-limb joint amplitudes | 18 weeks
  clinical evolution of lower-limb joint amplitudes using the modified Aschworth scale
compare the patients' mood evolution | 18 weeks
  patients' mood evolution using the Hospital Anxiety and Depression (HAD) scale
compare the evolution of cognitive disorders | 18 weeks
  evolution of cognitive disorders using the Cerebellar Cognitive Affective/Schmahmann Syndrome Scale (CCAS)
compare the before-after variation in the daily number of steps | 18 weeks
  before-after variation in the number of steps taken daily under ecological conditions, reported by pedometer
compare the before-after variation in heart rate | 18 weeks
  before-after variation in heart rate during walking assessments (6-minute and 10-meter tests)
compare the frequency and intensity of vesico-sphincter disorders | 18 weeks
  compare the frequency of vesico-sphincter disorders using Neurogenic Bowel Dysfunction sore
compare the anorectal disorders | 18 weeks
  compare the intensity of vesico-sphincter disorders using Urinary Symptom Profile
compare the quality of life | 18 weeks
  compare the quality of life using the EQ5D scale. The EQ-5D is a self-administered questionnaire that measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
compare the fatigue | 18 weeks
  compare the fatigue using the Modified Fatigue Impact Scale (MFIS)

CONTACTS AND LOCATIONS:
Locations (1):
- ICM, Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No